CLINICAL TRIAL: NCT02308553
Title: Phase I/II,Multicenter,Randomized,Double-blind,Placebo-controlled Trial Evaluating the Efficacy and Safety of Nintedanib/Vargatef in Combination With Paclitaxel Chemotherapy for Treatment of Patients With BRAF Wildtype Metastatic Melanoma
Brief Title: Efficacy and Safety of Nintedanib Combined With Paclitaxel Chemotherapy for Patients With BRAF wt Metastatic Melanoma
Acronym: NIPAWILMA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prof. Dr. med. Dirk Schadendorf (Other)
Collaborators: Boehringer Ingelheim (Industry); medac GmbH (Industry); Alcedis GmbH (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Dirk Schadendorf, Prof. Dr. med. Dirk Schadendorf, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nipawilma_2013
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cutaneous Malignant Melanoma
Keywords: BRAF V600 wildtype; cutaneous malignant melanoma; nintedanib; paclitaxel; kinase inhibitor
MeSH Terms: conditions — Melanoma, Cutaneous Malignant | interventions — nintedanib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nintedanib + Paclitaxel (Experimental): Nintedanib (150 or 200mg BID) for up to 48 weeks combined with paclitaxel 90mg/m2 BSA day 1, 8, 15 q28 days for a maximum of 6 courses
  Interventions: Drug: Nintedanib; Drug: Paclitaxel
- Nintedanib-Placebo + Paclitaxel (Placebo Comparator): Placebo (150 or 200mg BID) for up to 48 weeks combined with paclitaxel 90mg/m2 BSA day 1, 8, 15 q28 days for a maximum of 6 courses
  Interventions: Drug: Nintedanib-Placebo; Drug: Paclitaxel

INTERVENTIONS:
Drug: Nintedanib — Nintedanib (150 mg or 200 mg BID)
  Other Names: Vargatef
  Arms: Nintedanib + Paclitaxel
Drug: Nintedanib-Placebo — Placebo (150 mg or 200 mg BID)
  Arms: Nintedanib-Placebo + Paclitaxel
Drug: Paclitaxel — Paclitaxel as 90mg/mw infusion day 1, 8, 15 q28 (6 cycles)
  Other Names: Taxomedac

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase I/II trial designed to characterize the safety and estimate the efficacy of nintedanib when combined with paclitaxel chemotherapy compared with paclitaxel chemotherapy alone in patients with BRAF wild type metastatic melanoma not previously treated with taxanes or kinase inhibitors.

DETAILED DESCRIPTION:
Study Phase I: Run-In-Phase Based on acceptable safety data for nintedanib monotherapy, a rapid dose finding will be conducted in a classical 3+3 design. Predefined dose levels are 150 mg (dose level 1) and 200 mg (dose level 2) nintedanib, twice daily, with weekly paclitaxel 90 mg/m2.

Study Phase II Patients with advanced (unresectable Stage III or IV) BRaf V600 wild type melanoma (n=120) will be randomized (1:1) to receive either Nintedanib (150 or 200 mg BID depending on results of phase I) in combination with paclitaxel or Placebo in combination with paclitaxel.

Total study duration per patient: approximately 12 months of therapy + Follow up until end of study

All patients enrolled in either phase I or phase II will be treated according to the following treatment plan:

Week 1 - 24:

Chemotherapy with paclitaxel combined with nintedanib/placebo

Week 25 - 48:

Extended monotherapy with nintedanib/placebo

Week 52 (or approximately 4 weeks after last treatment dose):

End of Treatment visit

Follow up:

After end of treatment the survival, disease status and further therapies of each patient will be assessed every 3 months until death, progression of disease or end of study whichever occurs first

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, (surgically incurable or unresectable) stage III or IV, BRAF V600 wildtype metastatic cutaneous malignant melanoma.
2. Written informed consent
3. A minimum of 1 measurable lesion according to RECIST v1.1 criteria.
4. ECOG of 0-1.
5. Adequate hematologic, renal and liver function within 14 days prior to initiation of dosing:

   * Hematologic:

     * Absolute neutrophil count (ANC) ≥1.5 x 109/L
     * Hemoglobin ≥ 9 g/dL (5.6 mmol/L; Subjects may not have had a transfusion within 7 days of screening assessment)
     * Platelets: ≥ 100 x 109/L
   * Hepatic

     * Total bilirubin: ≤ 1.0 x ULN
     * AST and ALT: ≤ 1.5 x ULN (In the case of liver metastases: 2.5 x ULN)
   * Renal o Serum creatinine: ≤ 1.5 mg/dL (133 µmol/L) or, if greater than 1.5 mg/dL: Calculated creatinine clearance: ≥ 50 mL/min
6. effective method of contraception for at least 3 months after completion of nintedanib/placebo monotherapy as directed by their physician.
7. Men should use an effective method of contraception during treatment and for at least 6 months after completion of paclitaxel treatment and for at least 3 months after completion of nintedanib/placebo monotherapy as directed by their physician.
8. Patients must have recovered from all prior treatment-related toxicities to NCI CTCAE (v4.0) Grade of 0 or 1, except for toxicities not considered a safety risk such as alopecia.
9. Male or female, aged 18 years or older
10. Life expectancy at least 3 months

Exclusion Criteria:

1. Prior systemic therapy with taxanes or kinase inhibitors. Any prior therapy for metastatic disease must have been discontinued at least 4 weeks prior to initiation of dosing.
2. Major surgery or radiation therapy within 4 weeks of starting the study treatment (minor surgical procedures such as biopsies are allowed, however patients must have recovered).
3. Known inherited predisposition to bleeding or thrombosis and therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325mg per day)

   Patients with the following coagulation parameters will be excluded:
   * International normalised ratio (INR) > 2
   * Prothrombin time (PT) and partial thromboplastin time (PTT): > 50% of deviation of institutional ULN
4. History of clinically significant haemorrhagic or thromboembolic event in the past 6 months
5. NCI CTCAE (V4.0) grade 3 hemorrhage within 4 weeks of starting the study treatment.
6. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to randomization.
7. Serious, non-healing wound, ulcer, or bone fracture.
8. Known CNS disease:

   * Previous Grade 2 or higher sensory neuropathy.
   * History of or known spinal cord compression, or carcinomatous meningitis, or evidence of active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomization) or leptomeningeal disease on screening CT or MRI scan.
9. Any of the following within the 6 months prior to enrolment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
10. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
11. Ongoing cardiac dysrhythmias of NCI CTCAE Version 4.0 grade ≥ 2.
12. Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
13. Symptomatic peripheral vascular disease.
14. Proteinuria at screening as demonstrated by urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
15. Known hypersensitivity reaction to any of the components of study treatment (e.g. contrast media) or other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
16. Previous cancer (unless a RFS interval of at least 5 years) with the exception of surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin.
17. Known clinically uncontrolled infectious disease including HIV positivity or AIDS-related illness and active or chronic hepatitis C and/or B infection.
18. Pregnancy (absence to be confirmed by ß-hCG test) or lactation period.
19. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
20. Active alcohol or drug abuse
21. Treatment with other investigational drugs or treatments in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial.
22. Legal incapacity or limited legal capacity
23. Significant weight loss (> 10% of body weight) within past 6 months prior to inclusion into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 12 months after LPI
  Time from administration of first study drug to the date of first documented progression or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall survival | 12 months after LPI
  Time from the date of first administration of study drug to the date of death due to any cause.
Safety and toxicity (graded according to CTCAE, Version 4.0) | 12 months after LPI
  Reporting of adverse events from the date of first administration of study drug until 30 days after last administration of study drug
Quality of Life (EORTC QLQ-C30) | 12 months after LPI
  Quality of life during therapy (i.e. until end of treatment visit)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (10):
- Germany (10):
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - Elbeklinikum Buxtehude, Buxtehude
  - SRH Wald-Klinikum Gera, Gera
  - National Centre for Tumour Diseases (NCT), Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - University Hospital München, München
  - University Hospital Münster, Münster
  - Fachklinik Hornheide, Münster

IPD SHARING:
Plan to Share IPD: No